CLINICAL TRIAL: NCT02394886
Title: A Phase I Clinical Study to Evaluate the Safety of ALLO-ASC-DFU in the Patients With Diabetic Foot Ulcers
Brief Title: Safety of ALLO-ASC-DFU in the Patients With Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-ASC-DFU-101
Record Dates: First submitted 2015-03-03; First posted 2015-03-20 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALLO-ASC-DFU (Experimental): ALLO-ASC-DFU treatment with conventional care
  Interventions: Biological: ALLO-ASC-DFU

INTERVENTIONS:
Biological: ALLO-ASC-DFU

SUMMARY:
This is a phase I open-label study to evaluate the safety of ALLO-ASC-DFU in diabetic foot ulcers patients. ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide an new option in treating a diabetic foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 80 years of age.
2. Subject is diagnosed with Type I or Type II diabetes.
3. Subjects who have a wound defined as diabetic foot ulcer presence for more than 4 weeks, but not present for more than 54 weeks at the screening visit.
4. Foot ulcer located below the malleoli on plantar or dorsal surface of the foot and ulcer size is between 1 cm^2 and 25 cm^2.
5. Ulcer extends into the dermis or subcutaneous tissue without evidence of exposed muscle, tendon, bone, or joint capsule.
6. Ulcer is free of necrotic debris, exhibits no signs of clinical infection, and appears to be made of primarily vascularized tissue.
7. 0.7 < Ankle Brachial Index (ABI) < 1.3.
8. Subject is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Ulcer is of non-diabetic pathophysiology.
2. Gangrene is present on any part of the affected foot.
3. Ulcer is over an active Charcot deformity.
4. The ulcer has increased or decreased in size by 30% or more during one week after the screening visit.
5. The longest dimension of the Index Ulcer exceeds 5 cm at the screening visit.
6. Subject is Human Immunodeficiency Virus (HIV) positive.
7. Subjects with severe hepatic deficiencies.
8. Subjects with a glycated hemoglobin A1c (HbA1c) level of > 12%.
9. Subject who are allergic or have a hypersensitive reaction to bovine-derived proteins or fibrin glue.
10. Subjects requiring intravenous (IV) antibiotics to treat the index wound infection.
11. Subjects who are currently receiving dialysis.
12. Subjects who are pregnant or breast-feeding.
13. Subjects who are unwilling to use an "effective" method of contraception during the study.
14. Current evidence of osteomyelitis, cellulitis, or other evidence of infection including pus drainage from the wound site.
15. Subjects who have a clinically relevant history of alcohol or drugs abuse.
16. Subject's blood sugar is > 450 mg/dL at postprandial.
17. Subjects who are not able to understand the objective of this study or to comply with the study requirements.
18. Subjects who are considered to have a significant disease which can impact the study by the investigator.
19. Subjects who are considered not suitable for the study by the investigator.
20. Subjects who have a history of surgery for malignant tumor within the last five years (except carcinoma site).
21. Subjects who are currently or were enrolled in another clinical study within 60 days of screening.
22. Subjects who have undergone wound treatments with growth factors, dermal substitutes, or other biological therapies within the last 30 days.
23. Subjects who are receiving oral or parenteral corticosteroids, immunosuppressive, or cytotoxic agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 4 weeks

SECONDARY OUTCOMES:
Wound size and depth measurement | baseline and 1, 2, 4 weeks
  Evaluation of the improvement of wound measured by size and depth, and examines the change for 4 weeks period.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Pio Hong, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea